CLINICAL TRIAL: NCT03154138
Title: Assessment of the Rehabilitation of Postural Imbalance After Chronic Right Supratensorial Stroke by Prismatic Adaptation: Multicentric Randomised Sham-controlled Trial
Brief Title: Prismatic Adaptation for Rehabilitation of Postural Imbalance After Stroke
Acronym: PEQUIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Claude Bernard University (Other); Equipe " ImpAct Trajectoires " du Centre de Recherche en Neurosciences de Lyon (CRNL) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 69HCL17_0172
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Chronic Right Supratensorial Stroke Patients
Keywords: Stroke; hemiplegia; rehabilitation; prismatic adaptation; postural imbalance; posture; spatial cognition
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prismatic adaptation (PA) group (Experimental): Patients in the experimental group will benefit from 10 sessions of adaptation prismatic (PA) by means of one daily session of 20 minutes (5 times by week; 2 weeks), performed by an experienced physical therapist or occupational therapist. All patients will also benefit from conventional rehabilitation (Standard physical therapy, standard occupational therapy, standard speech therapy …) according to the needs of the patients.
  Interventions: Device: The prismatic adaptation (PA)
- Sham group (Placebo Comparator): Patients in the sham group will benefit from 10 sessions of sham adaptation prismatic (S-PA) by means of one daily session of 20 minutes (5 times by week; 2 weeks), performed by an experienced physical therapist or occupational therapist. All patients will also benefit from conventional rehabilitation (Standard physical therapy, standard occupational therapy, standard speech therapy …) according to the needs of the patients.
  Interventions: Device: The sham prismatic adaptation (S-PA)

INTERVENTIONS:
Device: The prismatic adaptation (PA) — Prismatic adaptation (PA) is based on the wearing of a pair of glasses producing a visual field deviation of 10° to rightward. While wearing theses glasses, the patient is asked to perform fast pointing movements towards targets by the right hand. Targets are symmetrical located at 10° in the right and left side in front of the patient. The order of pointing between these two targets is pseudo-randomly by the therapist. At the beginning of the exposure, the patient performs pointing movements with a shift toward the right side (initial errors consecutive to the prism deviation). Taking into account theses errors, the patient then compensates the optical deviation. After removing the prismatic glasses, the asked pointing movement to the targets is once again shifted but to the left side this time (after-effects attesting the prismatic adaptation)
  Arms: Prismatic adaptation (PA) group
Device: The sham prismatic adaptation (S-PA) — The sham prismatic adaptation (S-PA) is based on the wearing of a pair of glasses producing no visual field deviation. Theses sham glasses is identical with theses used in PA group without the optical deviation. The conditions are similar with theses in the PA group.
  The procedure with the sham glasses are similar with these one used in the PA group: While wearing the sham glasses, the patient is asked to perform fast pointing movements towards targets by the right hand. Targets are symmetrical located at 10° in the right and left side in front of the patient. The support with targets are the same as these one used in the PA group. The order of pointing between these two targets is pseudo-randomly by the therapist. At the beginning of the exposure, the patient performs pointing movements without shift. No compensation of movement is observed. After removing the prismatic glasses, the asked pointing movement to the targets is not shifted (No after-effects observed)
  Arms: Sham group

SUMMARY:
Postural imbalance after stroke leads to limitations of activity and a worse autonomy. The postural imbalance is increased in right supratensorial stroke (RSS) compared to left supratensorial stroke. The evidences for the rehabilitation of postural imbalance are weak.

Likewise, disorders of spatial reference frames are increased in RSS. The postural imbalance is correlated with the disorders of spatial reference frames in RSS patients.

Prismatic adaptation (PA) is often used for the rehabilitation of unilateral spatial neglect after RSS. Several studies have demonstrated a peculiar expansion of sensorimotor after-effects to spatial cognition. An immediate effect of reduction in postural imbalance have been showed in acute RSS. Therefore, it is interested to investigate the immediate and delayed effects of PA on the postural balance and the spatial reference frames in chronic RSS to purpose a new therapeutic approach.

The hypothesis of the study is that PA would improve the postural balance (activity) of chronic RSS patients by a reduction in mediolateral postural asymmetry, resulting from a " bottom-up " action of PA on spatial reference frames.

ELIGIBILITY:
Inclusion Criteria:

* Adult, over 18 years old, and less than 80 years old
* Stroke

  * right
  * supratensorial,
  * unilateral,
  * haemorrhagic or ischemic,
  * chronic (over 12 months)
* Ability to stay over 30 seconds in standing static position with open eyes and close eyes
* Show a postural imbalance, determined by a body weight bearing on right lower limb ≥ 60% during at least one posturographic evaluation with open eyes and that requires an inpatient rehabilitation
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research
* Free, enlightened and written consent of the patient

Exclusion Criteria:

* Cerebellar lesion
* Brainstem lesion
* Bilateral cerebral lesion
* All orthopaedic or rheumatologic diseases, retinal visual impairments or other diseases interfering with assessments in accordance with the investigator's judgment
* Pregnancy or breast feeding
* Under an administrative or legal supervision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Balance: The inter-group difference of within-group changes for the Berg Balance Scale (BBS) | Change from baseline (mean of the 2 pre-tests) at 7 days after the end of treatment (3 weeks about after the baseline)
  Balance : The inter-group difference of within-group changes for the Berg Balance Scale (BBS) Score between 0 and 56 points

SECONDARY OUTCOMES:
Balance: the inter-group difference of within-group changes for the Berg Balance Scale (BBS) | Change from baseline at 1 month after the end of treatment
  Change from baseline (mean of the 2 pre-tests) at one month after the end of treatment (M+1) (1 month and 2 weeks about after the baseline) and at three months after the end of treatment (M+3) (3 month and 2 weeks about after the baseline) Score between 0 and 56 points.
Balance: The inter-group difference of within-group changes for standing static posturographic variables | Change from baseline at +2 Hours, Day 3, Day7, Month +1 and Month +3 after the end of treatment
  Satnding posturographic variables include mediolateral and anteroposterior deviation of center of pression (COP), mediolateral and anteroposteriorvariability of COP, sway area of COP, body weight bearing on each lower limb.
  The mediolateral and anteroposterior deviations of COP measured in millimeters, the sway area of COP calculated in square millimeters, the mediolateral and anteroposterior variability of COP calculated as the standard deviation of the mediolateral and anteroposterior deviations of COP, body weight bearing on each lower limb measured in percent of total weight bearing.
Lateropulsion: The inter-group difference of within-group changes for the Scale for Contraversive Pushing (SCP) | Change from baseline at +2 Hours, Day 3, Day7, Month +1 and Month +3 after the end of treatment.
  Score between 0 and 6 points
The inter-group difference of within-group changes for each spatial reference frame (MSSA, VSSA, OLP, LBA) | Change from baseline at +2 Hours, Day 3, Day 7, Month 1 and Month 3 after the end of treatment
  Spatial reference frames include the measurement of the manual subjective straight aheaed (MSSA), the visual subjective straight ahead (VSSA), open-loup pointing without visual feedback (OLP), the subjective longitudinal body axis (LBA) Angular deviation measured in degrees
Autonomy : Inter-group difference of within-group changes for the Barthel index (BI) | Change from baseline (pre-test) at Day7, Month +1 and Month +3 after the end of treatment.
  Score between 0 and 100 points
Additionnal descriptive anatomic study of cerebral lesions using diffusion tensor Magnetic Resonance Imaginig (MRI) (Tractography) | Before the starting of the intervention, during the pre-tests.
  To determine the location of the cerebral lesion, the size of cerebral lesion and to quantify the severity of the disconnection (after tractography reconstructions of white matter pathways).
Relationship between prismatic adaptation induced changes on misperceptions of spatial reference frames and these on postural and balance disorders | +2Hours, Day+3, Day+7, Month+1 and Month+3.
  Statistical correlations between changes (before versus after intervention) on Berg Balance Scale (BBS), postural disorders (i.e. Weight Beainf Asymetry (WBA), body sway, and lateropulsion), and spatial reference frames.

CONTACTS AND LOCATIONS:
Overall Officials: Amandine GUINET-LACOSTE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - CHU Grenoble, Grenoble
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Henry Gabrielle, service de médecine physique et réadaptation, Saint-Genis-Laval

REFERENCES:
- [Derived] Hugues A, Guinet-Lacoste A, Bin S, Villeneuve L, Lunven M, Perennou D, Giraux P, Foncelle A, Rossetti Y, Jacquin-Courtois S, Luaute J, Rode G. Effects of prismatic adaptation on balance and postural disorders in patients with chronic right stroke: protocol for a multicentre double-blind randomised sham-controlled trial. BMJ Open. 2021 Nov 24;11(11):e052086. doi: 10.1136/bmjopen-2021-052086. PMID 34819284